CLINICAL TRIAL: NCT01136798
Title: Impact of Exenatide on Sleep and Circadian Function in Type 2 Diabetes: A Pilot Study
Brief Title: Impact of Exenatide on Sleep in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09-291-B
Record Dates: First submitted 2010-04-13; First posted 2010-06-03 (Estimated); Results first posted 2018-07-31 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-08

CONDITIONS: Type 2 Diabetes; Sleep Disordered Breathing
Keywords: slow wave sleep; exenatide and sleep
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Sleep Apnea Syndromes | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Usual T2 DM med regimen (Placebo Comparator): Subjects will continue on Type 2 DM therapy but will add placebo injected subcutaneously twice daily to their regimen for a total of 6 weeks.
  Interventions: Drug: Placebo
- Usual T2 DM med regimen plus Exenatide (Experimental): Subjects will continue on Type 2 DM therapy but will add injectable exenatide to their regimen There will be twice daily treatment with subcutaneous injections of 5 µg of Exenatide for 2 weeks followed by 4 weeks of treatment with twice daily subcutaneous injections of 10 µg of Exenatide.
  Interventions: Drug: Exenatide

INTERVENTIONS:
Drug: Exenatide — Exenatide or placebo medication administered subcutaneously 5 mcg twice daily for 2 weeks, followed by 10 mcg twice daily for 4 weeks
  Arms: Usual T2 DM med regimen plus Exenatide
Drug: Placebo — Exenatide or placebo medication administered subcutaneously 5 mcg twice daily for 2 weeks, followed by 10 mcg twice daily for 4 weeks
  Arms: Usual T2 DM med regimen

SUMMARY:
The investigators propose a pilot study to test the novel hypothesis that Exenatide treatment in patients with type 2 diabetes results in improved sleep duration and quality and to explore the relationship between improvements in sleep and measures of metabolic and circadian function. This project would be the first to probe the relationship between incretin hormone regulation, duration and intensity of sleep, glucose tolerance and circadian dysfunction in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of T2DM based on physician documentation according to established guidelines will be eligible.

Exclusion Criteria:

* Patients with unstable cardiac, neurological or psychiatric disease
* Women who are pregnant or report trying to get pregnant will be excluded.
* Patients treated for obstructive sleep apnea (OSA) will be excluded.
* Patients with established OSA will be included only if they have declined treatment of OSA.
* Patients with morbid obesity (BMI ≥ 40 gk/m2)
* Patients on insulin
* Patients already taking an incretin-based drug will not be included
* Patients with renal disease (creatinine clearance <30 ml/min), gastroparesis and history of pancreatitis will also be excluded based on known possible adverse medication side effects.
* Patients taking an insulin secretagogue will be excluded.
* Patients with Hemoglobin A1c values greater than or equal to 10 will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-06-01 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2016-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eve Van Cauter, PhD, Principal Investigator — University of Chicago
Locations (2):
- United States (2):
  - The University of Chicago, Chicago, Illinois
  - University of Chicago, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual T2 DM Med Regimen | Usual T2 DM Med Regimen Plus Exenatide
Started | 10 | 8
Completed | 10 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual T2 DM Med Regimen | Usual T2 DM Med Regimen Plus Exenatide | Total
Number analyzed (Participants) | 10 | 8 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (7.6) | 52.8 (8.6) | 56.2 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 2 | 2 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African-American | 5 | 7 | 12
  Non-Hispanic White | 4 | 0 | 4
  Hispanic | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Non-REM Slow Wave Sleep
Description: Total minutes of non-REM sleep was measured
Time Frame: baseline and after 6 weeks of treatment
Population: The Electronic Sleep Recordings for one participant in Usual T2 DM med regimen were corrupted and could not be analyzed. One participant in Usual T2 DM med regimen plus Exenatide had a very short sleep periods during the study and his data could not be interpreted, therefore this patient was excluded from the analysis.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Usual T2 DM Med Regimen | Usual T2 DM Med Regimen Plus Exenatide
Number analyzed (Participants) | 9 | 7
minutes
  Baseline | 47.3 (37.3) | 34.3 (34.4)
  At 6 week | 57.3 (38.1) | 41.4 (40.3)

2. Primary Outcome: Total Amount of Slow Wave Activity
Description: Total amount of slow wave activity during sleep derived from laboratory polysomnogram was measured
Time Frame: baseline and after 6 weeks of treatment
Population: The second primary outcome measure, slow-wave activity (SWA) was not collected.
Arm/Group | Usual T2 DM Med Regimen | Usual T2 DM Med Regimen Plus Exenatide
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Sleep Efficiency During Polysomnographic Recording
Description: Sleep efficiency will be calculated as total sleep time over total recording time.
Time Frame: baseline and after 6 weeks of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of total recording time
Arm/Group | Usual T2 DM Med Regimen | Usual T2 DM Med Regimen Plus Exenatide
Number analyzed (Participants) | 9 | 7
percentage of total recording time
  Baseline | 84.3 (6.8) | 85.3 (6.1)
  At 6 week | 83.8 (9.2) | 89.4 (5.4)

4. Secondary Outcome: Minutes of Wake After Sleep Onset During Sleep Recording
Description: total amount of time spent awake after sleep onset and before morning awakening will be calculated
Time Frame: baseline and after 6 weeks of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Usual T2 DM Med Regimen | Usual T2 DM Med Regimen Plus Exenatide
Number analyzed (Participants) | 9 | 7
minutes
  Baseline | 70.4 (33.1) | 56.6 (23)
  At 6 week | 52.3 (26.7) | 36.6 (18.7)

5. Secondary Outcome: Severity of Obstructive Sleep Apnea
Description: The apnea-hypopnea index (AHI) will be calculated from polysomnographic recordings. The minimum score for AHI is 0 (zero), corresponding to total absence of apnea or hypopnea. There is no theoretical maximum score although scores above 100 are very rarely observed. The lower the AHI value, the better. Higher AHI values correspond to greater severity of sleep apnea, a worse outcome. There are no subscales. We use continuous AHI values to measure severity of obstructive sleep apnea.
Time Frame: baseline and after 6 weeks of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual T2 DM Med Regimen | Usual T2 DM Med Regimen Plus Exenatide
Number analyzed (Participants) | 9 | 7
units on a scale
  Baseline | 15.9 (9.6) | 16.4 (10.9)
  At 6 week | 16.5 (11.4) | 10.9 (10.2)

6. Secondary Outcome: Mean 24-h Blood Glucose Levels
Description: Mean plasma levels of glucose will be calculated from samples collected across the 24-h cycle.
Time Frame: baseline and after 6 weeks of treatment
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Usual T2 DM Med Regimen | Usual T2 DM Med Regimen Plus Exenatide
Number analyzed (Participants) | 10 | 8
mg/dl
  Baseline | 134.4 (18.1) | 142.2 (37.5)
  At 6 week | 141.3 (22.1) | 136.1 (39.2)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Usual T2 DM Med Regimen | Usual T2 DM Med Regimen Plus Exenatide
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/8
Other Adverse Events (participants affected / at risk) | 0/10 | 0/8

LIMITATIONS AND CAVEATS:
When the investigators were unblinded in August 2016, a randomization error originating from the industry sponsor was identified, where only 8 participants were randomized to exenatide while 10 were randomized to placebo.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No